CLINICAL TRIAL: NCT04862754
Title: Effect of Interval Training on Arterial Stiffness in Women With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Taha, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T REC/012/003094.
Record Dates: First submitted 2021-01-12; First posted 2021-04-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Arterial Stiffness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interval training (Experimental): Aerobic interval training. It consisted of a modified interval cycle ergometer training program (3 days a week for 8 weeks). AIT consisted of 8 min warm up, followed by four times of 4-min intervals with HR at 80% of submaximal predetermined HR, with active phases of 3 min of cycling at 60% of submaximal predetermined HR. The exercise session was terminated by 5 min cool down
  Interventions: Other: interval training exercise
- medical treatment (No Intervention): hypertensive medication

INTERVENTIONS:
Other: interval training exercise — interval training exercise
  Arms: interval training

SUMMARY:
this study is aiming to assess the chronic effect of the interval training program on arterial stiffness in women with hypertension

ELIGIBILITY:
Inclusion Criteria:

* physically inactive
* BMI 30-40
* Stage 1 and 2 hypertension
* Elevated BP as systolic BP ≥130 mm Hg and/or diastolic BP ≥85 mm Hg measured at the brachial artery.

Exclusion Criteria:

* Medications known to affect weight or appetite
* Any disease associated with exercise intolerance.
* Women were taking hormone replacement therapy

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Central arterial stiffness measurements (Pulse Wave Velocity [PWV], augmentation index ) | two months
  Pulse wave analysis (PWA) of the women in the two groups: pre and post treatment for pulse wave velocity (PWV) and augmentation index(AIx)
  Pulse Wave Velocity [PWV], augmentation index (AIx @75HR) and resting heart rate were measured using analysis equipment which called Non-invasive blood pressure measurement system using "Mobil-O-Graph 24h PWA " with Hypertension Management Software Client Server (HMS-CS 4.3). PWA was performed using an oscillometric Mobil-O-Graph R 24 h PWA Monitor device (I.E.M GmbH, Germany) with integrated ARCSolver® software

SECONDARY OUTCOMES:
blood lipid profile | two months
  blood analysis will be used to measure lipid profile (high and low-density lipoprotein, cholesterol, triglyceride)
interleukin 6 | two months
  blood analysis will be used to measure interleukin 6
blood pressure (systolic and diastolic) | two months
  resting Blood pressure was monitored from the right arm using an automated digital electronic BP monitor (Omron digital BP monitor, Model 11 EM 403c; Tokyo Japan).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Egypt